CLINICAL TRIAL: NCT00428285
Title: A Phase II, Prospective, Open-label, Pilot Study of the Tolerability, Safety, and Efficacy of Argon Plasma Coagulation for the Treatment of Anal Intraepithelial Neoplasia Grade 2 or 3 in HIV-positive Men Having Sex With Men
Brief Title: Tolerability, Safety, & Efficacy of Argon Plasma Coagulation to Treat Anal Intraepithelial Neoplasia in HIV-Positive Men
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); CIHR Canadian HIV Trials Network (Network)
Responsible Party: Principal Investigator, Alexandra de Pokomandy, MD, Centre hospitalier de l'Université de Montréal (CHUM)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTN-216; SL06-0.11 (CHUM)
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Anus Neoplasms; HIV Infections
Keywords: Human Papilloma Virus; HIV infected MSM; Treatment Experienced; Treatment Naive; Anal Intraepithelial Neoplasia
MeSH Terms: conditions — Anus Neoplasms; HIV Infections | interventions — Argon Plasma Coagulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental)
  Interventions: Procedure: Argon Plasma Coagulation

INTERVENTIONS:
Procedure: Argon Plasma Coagulation — Argon Plasma Coagulation (APC) is a non-contact electrosurgical technique delivering a high-frequency electrical current through ionized argon gas i.e. the argon plasma. This current produces a zone of coagulation, desiccation, and devitalisation 2-3 mm deep. Patients will be offered up to 3 treatments if recurrence occur after the first two.

SUMMARY:
The purpose of this study is to assess if argon plasma coagulation (APC) is a safe and well tolerated treatment method for anal intraepithelial neoplasia (AIN) grade 2/3 in HIV-positive men having sex with men (MSM).

DETAILED DESCRIPTION:
HIV infected men having sex with men (MSM) are at increased risk of developing anal cancer compared to the general population and the incidence continues to increase despite better control of HIV infection with HAART (Highly Active Anti-Retroviral Therapy). The causative agent is known to be Human Papilloma Virus infection which can lead to dysplastic changes in the anus, detectable by High Resolution Anoscopy with biopsies. The analysis of the abnormal tissue can then be graded as Anal Intraepithelial Neoplasia 1 to 3, with AIN 2 or 3 considered as high grade dysplasia. These lesions are cancer precursors, but the proportion of lesions progressing to invasive anal cancer and the time to event are unknown. There is currently no recognized treatment to offer as standard of care although it is of general belief that treating these lesions, as it is done for women with CIN 2 and 3 (Cervical Intraepithelial Neoplasia) could help decrease the number of progressions to invasive anal cancer in MSM infected with HIV.

By experience at our center and results of this technique for other gastrointestinal pathologies, we believe Argon Plasma Coagulation (APC) could be a safe, well tolerated and efficient treatment of high-grade dysplasia (AIN 2/3) in HIV infected MSM.

This study will assess the APC treatment in 20 patients, all HIV infected MSM, with established AIN 2/3 (as confirmed with their last two anal biopsies, at least 4 months apart). Patients will then be followed with regular High Resolution Anoscopies for two years. The primary objective is to assess if APC is a safe and well tolerated treatment method for AIN 2/3 in HIV-positive MSM. As secondary objectives, the efficacy of APC treatment on AIN 2/3 lesions in HIV-positive MSM, the number of treatments with APC necessary to obtain regression or resolution of AIN 2/3 over two years and the efficacy of APC treatment to decrease anal HPV in this population will also be addressed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* The last two High Resolution Anoscopies (HRA) of the patient, occurring at least 4 months apart, revealed histologic diagnoses of AIN 2 or 3
* HIV infected for at least 6 months
* Patient must be a man having sex with other men (currently or anteriorly).
* Able to provide a signed and dated Research Ethics Board (REB)-approved informed consent form (ICF) for the study

Exclusion Criteria:

* History of invasive anal cancer
* International normalized ratio (INR) > 1.5
* Platelet count < 50,000
* Previously (or currently) received chemotherapy or radiotherapy for AIN or anal cancer
* Currently receiving interferon or cidofovir treatment
* Diagnosed with circumferential (diffuse) high-grade AIN, or involving > 75% of the anal canal.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-02; Primary Completion 2010-02 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
High grade dysplasia (AIN 2/3) | at 1 and 2 years

SECONDARY OUTCOMES:
Anal human papilloma virus (HPV) | at 1 and 2 years
Tolerability and safety of the treatment | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra de Pokomandy, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM); George Ghattas, MD, Principal Investigator — McGill University Health Center and Centre Hospitalier de l'Université de Montréal (CHUM)
Locations (2):
- Canada (2):
  - Notre-Dame Hospital (Centre Hospitalier de l'Université de Montréal), Montreal, Quebec
  - Royal Victoria Hospital (McGill University Health Center), Montreal, Quebec

REFERENCES:
- [Result] de Pokomandy A, Rouleau D, Lalonde R, Beauvais C, de Castro C, Coutlee F; Human Immunodeficiency and Papilloma Virus Research Group (HIPVIRG) Study Group. Argon plasma coagulation treatment of anal high-grade squamous intraepithelial lesions in men who have sex with men living with HIV: results of a 2-year prospective pilot study. HIV Med. 2018 Feb;19(2):81-89. doi: 10.1111/hiv.12544. Epub 2017 Aug 23. PMID 28833949